CLINICAL TRIAL: NCT02693379
Title: Cervical Cancer Screening in Madagascar: Usability of Mobile Telemedicine for Detection of Precancerous Lesions From Smartphone Photos
Brief Title: Cervical Cancer Screening in Madagascar Using Smartphone Photos and Mobile Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Patrick Petignat (Other)
Responsible Party: Sponsor-Investigator, Prof. Patrick Petignat, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-071
Record Dates: First submitted 2015-07-08; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Cervical Precancer
Keywords: cervical cancer; HPV; VIA; screening; smartphone; telemedicine
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- D-VIA (Experimental): HPV high risk-positive (16, 18, 45, 31, 33, 35, 39, 51, 52, 56, 58, 59, 66, 68) women had a cervical examination using acetic acid (VIA) application and visual inspection.
  Interventions: Device: D-VIA

INTERVENTIONS:
Device: D-VIA — D-VIA images were captured during the cervical examination with a smartphone. Biopsies and cytological samples were taken on all patients and analyzed for gold standard results. Images were shown to off site experts. D-VIA and VIA diagnoses were then compared.
  Women who were diagnosed on-site as pathological underwent appropriate treatment at the same consultation. Women who were diagnosed as pathological later by histopathological analyses were asked to return to the clinic for treatment.

SUMMARY:
The purpose of this study is to determine whether smartphone photos may assist health-care worker (on-site) and to evaluate the diagnostic reliability and accuracy of cervical examination with smartphone photos of VIA (D-VIA), on-site and off-site, compared with conventional VIA, for human papillomavirus (HPV) positive women.

DETAILED DESCRIPTION:
Background: Cervical cancer is the leading cause of cancer death in females in Madagascar. In this country, a large-scale screening of precancerous lesions with cytology is hardly possible, because of the lack of specialists and infrastructures. Visual inspection of the cervix with application of 5% acetic acid (VIA) is an inexpensive alternative but very subjective since it depends on the examiner's experience. Mobile telemedicine is a very promising tool in order to assist non-expert health-care workers in rural area for cervical cancer screening.

Objective: To assess if Smartphone may assist health-care worker (on-site) and to evaluate the diagnostic reliability and accuracy of cervical examination with smartphone photos of VIA (D-VIA) compared with conventional VIA, for women testing positive for human papillomavirus (HPV).

Material and method: On-site health care workers will be trained in VIA. Prescreened HPV-positive women will be referred to VIA evaluation, during which digital images with a smartphone (D-VIA) will be taken for later evaluation by a VIA specialist in Geneva linked by telemedicine. Women with positive VIA results will be treated with cold coagulation if eligible. Histological results will be considered as gold standard. The results will be analyzed with Cohen's kappa coefficient, Mcnemar's test and Bonferroni's adjustment for multiple comparisons to assess the performance of D-VIA.

Expected results: Based on the results of this project, the investigators will develop an educational training and quality assurance program for health providers for VIA and so contribute to a scaling-up of cervical cancer control. An appropriate triage by VIA will reduce not only an excessive referral rate but also an excessive treatment delay, giving the possibility of a "screen (HPV), see (VIA/D-VIA), and treat" program in a single or two visits.

ELIGIBILITY:
Inclusion Criteria:

* 30-49 years
* HPV-positive
* Attending the cervical cancer screening program conducted by the Saint-Damien Health-Care Centre
* Understands study procedures and accepts voluntarily to participate by signing the informed consent form (ICF)

Exclusion Criteria:

* Previous Hysterectomy
* Conditions that can interfere with visualization of the cervix
* Pregnancy > 20 weeks
* Not able to comply with protocol study.

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1041 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Differences in sensitivity and specificity of VIA examination (control) and digital VIA to detect cervical cancer and pre-cancer | up to 12 months
  Sensitivity and specificity will be calculated using histological results as gold-standard. All lesion Cin2 and worse will be considered as pathological.

SECONDARY OUTCOMES:
Overall agreement between diagnoses based on VIA examination (control) and diagnoses for the same patient based on digital VIA. | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Petignat, Professor, Principal Investigator — University Hospital, Geneva
Locations (1):
- Saint-Damien Health-Care Centre, Ambanja, Antsiranana, Madagascar

IPD SHARING:
Plan to Share IPD: Yes
Data will be used for scientific publications and congress presentations.

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Marquardt K. [Correlation of cervical cytology and histology]. Pathologe. 2011 Nov;32(6):491-6. doi: 10.1007/s00292-011-1479-2. German. PMID 21822676
- See also: Health Profile Madagascar. World Life Expectancy. Last time accessed: 15.01.2014 — http://www.worldlifeexpectancy.com/country-health-profile/madagascar
- See also: WHO/ICO. Information Centre on HPV and Cervical Cancer (HPV Information Centre) - Human Papillomavirus and Related Cancers in Madagascar. Summary Report 2010. 2010. — http://www.hpvcentre.net/statistics/reports/XWX.pdf